CLINICAL TRIAL: NCT06792006
Title: Awareness Assessment of Climate Change Impacts Among a Group of University Students: a Cross-Sectional Study
Brief Title: Awareness of Climate Change Impacts Among University Students
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Samaa Sayed, Lecturer at Pediatric Dentistry and Dental Public Health Department, Cairo University, Cairo University
Other Study IDs: OMED121
Record Dates: First submitted 2025-01-14; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Climate Change
Keywords: climate change, College students, Awareness

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study evaluates college students' awareness of climate change and its effects on the environment through a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* All the university students are eligible to participate in the study

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: University students from various years of study
Sampling Method: Probability Sample
Enrollment: 273 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Assessment of the climate change awareness among a group of university students | through study competition, average one year
  The assessment of the climate change awareness among a group of university students will be done using a Validated questionnaire ( De Paula Baer, et al., 2019). Measuring unit will be percentage

IPD SHARING:
Plan to Share IPD: Undecided